CLINICAL TRIAL: NCT05284851
Title: A Random, Double-Blind, Multicenter, Positive Control and Placebo Control Phase Two Trail to Evaluate the Safety and Immunogenicity of Live Attenuated Influenza Vaccine in 3-59y Healthy People
Brief Title: The Safety and Immunogenicity Evaluation of Live Attenuated Influenza Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Collaborators: He Bei province Center for Disease control and prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Bchtpharm
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Influenza Prevention
Keywords: Immunogenicity; Safety; Live Attenuated Influenza Vaccine

STUDY DESIGN:
Intervention Model Description: Totally 2520 health people aged 3-59 years old will be divided into two age group, containing 1260 in 18-59 years old and 1260 in 3-19 years old. All subjects will receive vaccination either LAVI(non freeze- dried), LAVI(freeze- dried) or placebo in a ratio of 2:2:1.
Who Masked: Participant
Masking Description: The design of this trail is based on random, one-blind, placebo control. The subjects will not know the masking status, unless the specific subjects who required treatment for serious adverse events .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): Healthy people in experimental group will receive a dose of Live Attenuated Influenza Vaccine (non freeze- dried)
  Interventions: Biological: Live Attenuated Influenza Vaccine(non freeze-dried)
- Positive control group (Active Comparator): Healthy people in Positive control group will receive a dose of Live Attenuated Influenza Vaccine ( freeze- dried)
  Interventions: Biological: Live Attenuated Influenza Vaccine(freeze-dried)
- Placebo group (Placebo Comparator): Healthy people in placebo group will receive a dose of placebo
  Interventions: Biological: Live Attenuated Influenza Vaccine placebo

INTERVENTIONS:
Biological: Live Attenuated Influenza Vaccine(non freeze-dried) — Live Attenuated Influenza Vaccine Live Attenuated Influenza Vaccine placebo, containing H1, H3 and B type influenza Live Attenuated virus.
  Arms: Experimental group 1
Biological: Live Attenuated Influenza Vaccine(freeze-dried) — Live Attenuated Influenza Vaccine Live Attenuated Influenza Vaccine placebo, containing H1, H3 and B type influenza Live Attenuated virus.
  Arms: Positive control group
Biological: Live Attenuated Influenza Vaccine placebo — Live Attenuated Influenza Vaccine placebo, not containing H1, H3 and B type influenza Live Attenuated virus.
  Arms: Placebo group

SUMMARY:
Live Attenuated freeze-dried Influenza Vaccine has been licensed for use in 2020 (Approval No.S20200002), the sponsor of this research submitted an new application for non freeze-dried Live Attenuated Influenza Vaccine in 2021. The main objective of phase two trail is to evaluate the immunogenicity of LAVI (non freeze- dried). The secondary objective is to evaluate the safety of LAVI (non freeze- dried).

DETAILED DESCRIPTION:
Totally 2520 health people aged 3-59 years old will be divided into two age group, containing 1260 in 18-59 years old and 1260 in 3-19 years old. All subjects will receive vaccination either LAVI(non freeze- dried), LAVI(freeze- dried) or placebo in a ratio of 2:2:1.

All subjects will be collected any adverse events within 30 days and any serious adverse events within 6 months for safety evaluation. All subjects will be collected blood sample and nasopharyngeal swab for immunogenicity evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged in 3-59 years old
* Had not received vaccination of Influenza vaccine in the past one year
* Had not infected with Influenza virus
* This trail has been agreed by volunteers or his/her legal guardian
* Volunteers or his/her legal guardian will fellow this trail protocol

Exclusion Criteria:

* People with fever before vaccination, temperature higher than 37.0 #
* Females in suckling period, pregnancy (pregnancy test positive) or prepared to be pregnant
* People given whole blood, plasma or immunoglobulin therapy within 3 months before vaccination
* According to judgement of researchers, the subjects have any other factors that are not appropriate for this clinical trials
* Acute infectious disease or acute attack of chronic disease before inoculation
* People get any vaccine within 14 days before the trial
* People in immune deficiency or diagnosed with congenital or acquired immunodeficiency, people with immunosuppressive therapy in the past six months
* People with epilepsy or a history of mental illness

Ages: 3 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2520 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
The number of participants with positive sIgA as assessed by SAS v9.4 | within 10 days after vaccination
  The Mucosal convention rate of sIgA in all subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Provincial Center for Disease Control and Prevention, Shijiazhuang, Hebei, China